CLINICAL TRIAL: NCT02908100
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of GDC-0853 in Patients With Moderate to Severe Active Systemic Lupus Erythematosus
Brief Title: A Study of the Safety and Efficacy of GDC-0853 in Participants With Moderate to Severe Active Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA30044; 2016-001039-11 (EudraCT Number)
Record Dates: First submitted 2016-09-14; First posted 2016-09-20 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — fenebrutinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants received matching placebo to GDC-0853 orally starting on Day 1 and ending at Week 48, in combination with background standard of care therapy.
  Interventions: Drug: Placebo
- GDC-0853 (150mg) QD (Experimental): Participants received GDC-0853 (150mg) orally once daily (QD) starting on Day 1 and ending at Week 48, in combination with background standard of care therapy.
  Interventions: Drug: GDC-0853
- GDC-0853 (200mg) BID (Experimental): Participants received GDC-0853 (200mg) orally twice daily (BID) starting on Day 1 and ending at Week 48, in combination with background standard of care therapy.
  Interventions: Drug: GDC-0853

INTERVENTIONS:
Drug: GDC-0853 — Participants received GDC-0853 at dosages of 150 or 200mg as per the dosing schedules described above.
  Other Names: RO7010939
  Arms: GDC-0853 (150mg) QD; GDC-0853 (200mg) BID
Drug: Placebo — Participants received matching placebo to GDC-0853 at dosages of 150 and 200mg as per the dosing schedules described above.
  Arms: Placebo

SUMMARY:
This is a study to evaluate the safety and efficacy of GDC-0853 in combination with standard of care therapy in participants with moderate to severe active systemic lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of SLE classification criteria according to either American College of Rheumatology (ACR) or Systemic Lupus International Collaborating Clinics (SLICC) criteria at any time prior to or at screening
* At least one serologic marker of SLE at screening as follows: positive antinuclear antibody (ANA) test by immunofluorescent assay with titer >/= 1:80; or positive anti-double-stranded DNA (anti-dsDNA) antibodies; or positive anti-Smith antibody
* At both screening and Day 1, moderate to severe active SLE, defined as meeting all of the following unless indicated otherwise: Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score ≥ 8 (at screening only) with clinical SLEDAI-2K score >/= 4.0 (at both screening and Day 1), Physician's Global Assessment >/= 1.0 (out of 3), and currently receiving at least one standard oral treatment for SLE
* If on oral corticosteroids (OCS), the dose must be </= 40 mg/day prednisone (or equivalent)
* Stable doses of anti-malarial or immunosuppressive therapies
* Participants must be willing to avoid pregnancy

Exclusion Criteria:

* Proteinuria > 3.5 g/24 h or equivalent using urine protein-to-creatinine ratio (uPCR) in a first morning void urine sample
* Active proliferative lupus nephritis (as assessed by the investigator) or histological evidence of active Class III or Class IV lupus nephritis on renal biopsy performed in the 6 months prior to screening (or during the screening period)
* History of having required hemodialysis or high dose corticosteroids (>100 mg/d) prednisone or equivalent) for the management of lupus renal disease within 90 days of Day 1
* Neuropsychiatric or central nervous system lupus manifestations
* Serum creatinine > 2.5 mg/dL, or estimated glomerular-filtration rate < 30 milliliter per minute (mL/min) or on chronic renal replacement therapy
* History of receiving a solid organ transplant
* Evidence of active, latent, or inadequately treated infection with Mycobacterium tuberculosis (TB)
* Significant and uncontrolled medical disease within the 12 weeks prior to screening in any organ system (e.g., cardiac, neurologic, pulmonary, renal, hepatic, endocrine, metabolic, gastrointestinal, or psychiatric) not related to SLE, which, in the investigator's or Sponsor's opinion, would preclude study participation
* History of cancer, including hematological malignancy and solid tumors, within 10 years of screening
* Need for systemic anticoagulation with warfarin, other oral or injectable anticoagulants, or anti-platelet agents
* Evidence of chronic and/or active hepatitis B or C

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (69):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Valerius Medical Group & Research Ctr of Greater Long Beach, Los Alamitos, California
  - RASF-Clinical Research Center, Boca Raton, Florida
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Omega Research Consultants, Orlando, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Via Christi Research, a division of Via Christi Hospitals Wichita, Inc., Wichita, Kansas
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - The Arthritis & Diabetes Clinic, Inc.; Research, Monroe, Louisiana
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Saint Lawrence Health System, Canton, New York
  - New York University School of Medicine, New York, New York
  - Shanahan Rheumatology & Immunology, PLLC, Raleigh, North Carolina
  - Ohio State University Clinical Trials Management Office, Columbus, Ohio
  - Tekton Research Inc, Austin, Texas
  - Accurate Clinical Research, Houston, Texas
  - Arthritis Clinic Of Central Texas, San Marcos, Texas
- Argentina (5):
  - Organizacion Medica de Investigacion, Buenos Aires
  - APRILLUS, Buenos Aires
  - Hospital Italiano de La Plata, La Plata
  - CER San Juan Centro Polivalente de Asistencia e Investigacion Clinica, San Juan
  - Centro Medico Privado de Reumatologia; Reumathology, San Miguel
- Brazil (11):
  - CEDOES - Diagnóstico e Pesquisa, Vitória, Espírito Santo
  - CIP - Centro Internacional de Pesquisa X; Pesquisa Clinica, Goiânia, Goiás
  - Hospital das Clinicas - UFMG, Belo Horizonte, Minas Gerais
  - CMiP - Centro Mineiro de Pesquisa*X*, Juiz de Fora, Minas Gerais
  - Edumed - Educação e Saúde SA, Curitiba, Paraná
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas em Diabetes - CPD, Porto Alegre, Rio Grande do Sul
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - Hospital Estadual Mario Covas, Santo André, São Paulo
  - Hospital Abreu Sodré - AACD, São Paulo, São Paulo
- Bulgaria (6):
  - MHAT Plovdiv, Plovdiv
  - Medical Center "Teodora", EOOD, Rousse
  - Medical Center Excelsior OOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - MC "Synexus - Sofia", EOOD, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
- Chile (5):
  - CTR Estudios SPA, Providencia
  - Dermacross, Santiago
  - Centro de Estudios Reumatológicos, Santiago
  - SOMEAL, Santiago
  - Biomedica, Santiago
- Colombia (6):
  - CEQUIN - Fundación Cardiomet Eje Cafetero, Armenia
  - Centro Integral de Reumatologia del Caribe SAS CIRCARIBE SAS, Barranquilla
  - Centro de Reumatologia y Ortopedia, Barranquilla
  - Medicity S.A.S., Bucaramanga
  - Servimed S.A.S., Bucaramanga
  - Hospital Pablo Tobon Uribe, Medellín
- Charite Research Organisation GmbH; Phase - I Unit of Hematology and Oncology, Berlin, Germany
- Mexico (6):
  - Centro de Investigacion Alberto Bazzoni S.A. de C.V., Torreón, Coahuila
  - Unidad de Atencion Medica e Investigacion en Salud S.C., Mérida, Yucatán
  - Consultorio Particular del Dr. Miguel Cortes Hernandez, Cuernavaca
  - Hospital Angeles Lindavista, México
  - Hospital Universitario de Saltillo, Saltillo
  - Hospital Central Dr Ignacio Morones Prieto, San Luis Potosí City
- South Korea (2):
  - Konkuk University Medical Center, Seoul
  - The Catholic University of Korea St.Mary's Hospital, Seoul
- Spain (4):
  - Complejo Hospitalario Universitario A Coruña, A Coruña, LA Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico Universitario de Valladolid; Servicio de Reumatologia, Valladolid
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District
- United Kingdom (2):
  - University College London Hospital, London
  - Guy's Hospital; Louise Coote Lupus Unit, London

REFERENCES:
- [Derived] Isenberg D, Furie R, Jones NS, Guibord P, Galanter J, Lee C, McGregor A, Toth B, Rae J, Hwang O, Desai R, Lokku A, Ramamoorthi N, Hackney JA, Miranda P, de Souza VA, Jaller-Raad JJ, Maura Fernandes A, Garcia Salinas R, Chinn LW, Townsend MJ, Morimoto AM, Tuckwell K. Efficacy, Safety, and Pharmacodynamic Effects of the Bruton's Tyrosine Kinase Inhibitor Fenebrutinib (GDC-0853) in Systemic Lupus Erythematosus: Results of a Phase II, Randomized, Double-Blind, Placebo-Controlled Trial. Arthritis Rheumatol. 2021 Oct;73(10):1835-1846. doi: 10.1002/art.41811. Epub 2021 Aug 24. PMID 34042314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 69 centers in 12 countries.
Pre-assignment Details: An overall total of 616 participants were screened into the study, of which 356 participants were screen failures. 260 participants (Intent-To-Treat/ITT population) were randomized into the study, of which 1 participant did not receive any study treatment meaning that the Safety population consisted of 259 participants.
Period: Overall Study
Arm/Group | Placebo | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID
Started | 86 | 87 | 87
Completed | 63 | 66 | 66
Not Completed | 23 | 21 | 21
Not completed — Adverse Event | 7 | 6 | 9
Not completed — Death | 2 | 0 | 0
Not completed — Lack of Efficacy | 2 | 3 | 3
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Non-Compliance With Study Drug | 1 | 1 | 2
Not completed — Non-Compliance With Contraceptive Method | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Pregnancy | 1 | 2 | 0
Not completed — Withdrawal by Subject | 8 | 7 | 5
Not completed — Randomised in Error | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID | Total
Number analyzed (Participants) | 86 | 87 | 87 | 260
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (11.5) | 43.3 (12.4) | 40.4 (10.6) | 41.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 82 | 84 | 251
  Male | 1 | 5 | 3 | 9
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 54 | 61 | 61 | 176
    Not Hispanic or Latino | 32 | 25 | 26 | 83
    Not Stated | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    American Indian or Alaska native | 11 | 8 | 17 | 36
    Asian | 7 | 1 | 2 | 10
    Black or African American | 11 | 15 | 13 | 39
    Multiple | 1 | 1 | 3 | 5
    White | 56 | 62 | 52 | 170

OUTCOME MEASURES:

1. Primary Outcome: Systemic Lupus Erythematosus Responder Index (SRI)-4 Response at Week 48
Description: The Systemic Lupus Erythematosus Responder Index (SRI)-4 measures reduction in SLE disease activity and is a composite measure that includes the SLE Disease Activity Index (SLEDAI-2K), British Isles Lupus Activity Group (BILAG) 2004 and Physician Global Assessment. It is defined as: 1) Reduction of ≥4 points from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score; 2) no new British Isles Lupus Assessment Group (BILAG) A or no more than 1 new BILAG B disease activity scores and 3) no worsening (defined as an increase of ≥0.3 points [10 mm] from baseline) in the Physician's Global Assessment of Disease Activity. The score range is from 0 to 100, with higher scores indicating greater disease activity.
Time Frame: Week 48
Population: The Intent-To-Treat (ITT) population was defined as all randomized participants regardless of whether they received any study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID
Number analyzed (Participants) | 86 | 87 | 87
Percentage of Participants | 44.2 | 50.6 | 51.7
Statistical Analysis 1: Comparison: Placebo vs GDC-0853 (150mg) QD; Test type: Superiority; p = 0.373, Cochran-Mantel-Haenszel; Absolute Difference = 6.4, 95% CI 2-sided [-8.5 to 21.2]
Statistical Analysis 2: Comparison: Placebo vs GDC-0853 (200mg) BID; Test type: Superiority; p = 0.339, Cochran-Mantel-Haenszel; Absolute Difference = 7.5, 95% CI 2-sided [-7.3 to 22.4]

2. Secondary Outcome: SRI-4 Response at Week 48 With a Sustained Reduction of Oral Corticosteroids (OCS) Dose to Less Than (<)10 Milligrams Per Day (mg/Day) and Less Than or Equal to (</=) Day 1 Dose During Week 36 Through Week 48
Description: The SRI-4 measures reduction in SLE disease activity and is a composite measure that includes the SLE Disease Activity Index (SLEDAI-2K), British Isles Lupus Activity Group (BILAG) 2004 and Physician Global Assessment. It is defined as: 1) Reduction of ≥4 points from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score; 2) no new British Isles Lupus Assessment Group (BILAG) A or no more than 1 new BILAG B disease activity scores and 3) no worsening (defined as an increase of ≥0.3 points [10 mm] from baseline) in the Physician's Global Assessment of Disease Activity. The score range is from 0 to 100, with higher scores indicating greater disease activity. OCS tapering requires a sustained reduction of OCS from Week 36 through Week 48 [less than 10 milligram per day (mg/day) and less or equal to the dose received on Day 1].
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID
Number analyzed (Participants) | 86 | 87 | 87
Percentage of Participants | 41.9 | 50.6 | 44.8
Statistical Analysis 1: Comparison: Placebo vs GDC-0853 (150mg) QD; Test type: Superiority; p = 0.223, Cochran-Mantel-Haenszel; Absolute Difference = 8.7, 95% CI 2-sided [-6.1 to 23.5]
Statistical Analysis 2: Comparison: Placebo vs GDC-0853 (200mg) BID; Test type: Superiority; p = 0.737, Cochran-Mantel-Haenszel; Absolute Difference = 3.0, 95% CI 2-sided [-11.8 to 17.7]

3. Secondary Outcome: SRI-4 Response at Week 24 With a Sustained Reduction of OCS Dose to < 10 mg/Day and </= Day 1 Dose During Week 12 Through Week 24
Description: The SRI-4 measures reduction in SLE disease activity and is a composite measure that includes the SLE Disease Activity Index (SLEDAI-2K), British Isles Lupus Activity Group (BILAG) 2004 and Physician Global Assessment. It is defined as: 1) Reduction of ≥4 points from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score; 2) no new British Isles Lupus Assessment Group (BILAG) A or no more than 1 new BILAG B disease activity scores and 3) no worsening (defined as an increase of ≥0.3 points [10 mm] from baseline) in the Physician's Global Assessment of Disease Activity. The score range is from 0 to 100, with higher scores indicating greater disease activity. OCS tapering requires a sustained reduction of OCS from Week 12 through Week 24 [less than 10 milligram per day (mg/day) and less or equal to the dose received on Day 1].
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID
Number analyzed (Participants) | 86 | 87 | 87
Percentage of Participants | 43.0 | 47.1 | 47.1
Statistical Analysis 1: Comparison: Placebo vs GDC-0853 (150mg) QD; Test type: Superiority; p = 0.614, Cochran-Mantel-Haenszel; Absolute Difference = 4.1, 95% CI 2-sided [-10.7 to 18.9]
Statistical Analysis 2: Comparison: Placebo vs GDC-0853 (200mg) BID; Test type: Superiority; p = 0.607, Cochran-Mantel-Haenszel; Absolute Difference = 4.1, 95% CI 2-sided [-10.7 to 18.9]

4. Secondary Outcome: SRI-4 Response at Week 24
Description: The SRI-4 measures reduction in SLE disease activity and is a composite measure that includes the SLE Disease Activity Index (SLEDAI-2K), British Isles Lupus Activity Group (BILAG) 2004 and Physician Global Assessment. It is defined as: 1) Reduction of ≥4 points from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score; 2) no new British Isles Lupus Assessment Group (BILAG) A or no more than 1 new BILAG B disease activity scores and 3) no worsening (defined as an increase of ≥0.3 points [10 mm] from baseline) in the Physician's Global Assessment of Disease Activity. The score range is from 0 to 100, with higher scores indicating greater disease activity.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID
Number analyzed (Participants) | 86 | 87 | 87
Percentage of Participants | 46.5 | 52.9 | 52.9
Statistical Analysis 1: Comparison: Placebo vs GDC-0853 (150mg) QD; Test type: Superiority; p = 0.410, Cochran-Mantel-Haenszel; Absolute Difference = 6.4, 95% CI 2-sided [-8.5 to 21.2]
Statistical Analysis 2: Comparison: Placebo vs GDC-0853 (200mg) BID; Test type: Superiority; p = 0.418, Cochran-Mantel-Haenszel; Absolute Difference = 6.4, 95% CI 2-sided [-8.5 to 21.2]

5. Secondary Outcome: SRI-4 Response at Week 48 in Patients With High vs. Low Plasmablast Signature Levels
Description: The SRI-4 measures reduction in SLE disease activity and is a composite measure that includes the SLE Disease Activity Index (SLEDAI-2K), British Isles Lupus Activity Group (BILAG) 2004 and Physician Global Assessment. It is defined as: 1) Reduction of ≥4 points from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score; 2) no new British Isles Lupus Assessment Group (BILAG) A or no more than 1 new BILAG B disease activity scores and 3) no worsening (defined as an increase of ≥0.3 points [10 mm] from baseline) in the Physician's Global Assessment of Disease Activity. The score range is from 0 to 100, with higher scores indicating greater disease activity. The Plasmablast Signature (PB) is a Bruton's Tyrosine Kinase (BTK)-dependent blood RNA signature comprised of three genes (IgJ, MZB1 and TXNDC5). Q1/2/3/4 = Quartile 1/2/3/4.
Time Frame: Week 48
Population: The Intent-To-Treat (ITT) population was defined as all randomized participants regardless of whether they received any study drug. Data presented below is only for participants that were included in the actual analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID
Number analyzed (Participants) | 24 | 24 | 25
Percentage of Participants
  Plasmablast Signature Level Q1: number analyzed (Participants) | 24 | 21 | 20
  Plasmablast Signature Level Q1 | 37.5 | 52.4 | 45.0
  Plasmablast Signature Level Q2: number analyzed (Participants) | 22 | 24 | 19
  Plasmablast Signature Level Q2 | 54.5 | 54.2 | 63.2
  Plasmablast Signature Level Q3: number analyzed (Participants) | 19 | 21 | 25
  Plasmablast Signature Level Q3 | 36.8 | 52.4 | 52.0
  Plasmablast Signature Level Q4: number analyzed (Participants) | 20 | 21 | 23
  Plasmablast Signature Level Q4 | 50.0 | 42.9 | 47.8
Statistical Analysis 1: Comparison: Placebo vs GDC-0853 (150mg) QD; Plasmablast Signature Level Q1; Test type: Superiority; p = 0.378, Cochran-Mantel-Haenszel; Absolute Difference = 14.9, 95% CI 2-sided [-14 to 43.7]
Statistical Analysis 2: Comparison: Placebo vs GDC-0853 (200mg) BID; Plasmablast Signature Level Q1; Test type: Superiority; p = 0.732, Cochran-Mantel-Haenszel; Absolute Difference = 7.5, 95% CI 2-sided [-21.7 to 36.7]
Statistical Analysis 3: Comparison: Placebo vs GDC-0853 (150mg) QD; Plasmablast Signature Level Q2; Test type: Superiority; p = 0.500, Cochran-Mantel-Haenszel; Absolute Difference = -0.4, 95% CI 2-sided [-29.2 to 28.4]
Statistical Analysis 4: Comparison: Placebo vs GDC-0853 (200mg) BID; Plasmablast Signature Level Q2; Test type: Superiority; p = 0.234, Cochran-Mantel-Haenszel; Absolute Difference = 8.6, 95% CI 2-sided [-21.4 to 38.7]
Statistical Analysis 5: Comparison: Placebo vs GDC-0853 (150mg) QD; Plasmablast Signature Level Q3; Test type: Superiority; p = 0.364, Cochran-Mantel-Haenszel; Absolute Difference = 15.5, 95% CI 2-sided [-14.9 to 46]
Statistical Analysis 6: Comparison: Placebo vs GDC-0853 (200mg) BID; Plasmablast Signature Level Q3; Test type: Superiority; p = 0.134, Cochran-Mantel-Haenszel; Absolute Difference = 15.2, 95% CI 2-sided [-14.1 to 44.4]
Statistical Analysis 7: Comparison: Placebo vs GDC-0853 (150mg) QD; Plasmablast Signature Level Q4; Test type: Superiority; p = 0.830, Cochran-Mantel-Haenszel; Absolute Difference = -7.1, 95% CI 2-sided [-37.6 to 23.3]
Statistical Analysis 8: Comparison: Placebo vs GDC-0853 (200mg) BID; Plasmablast Signature Level Q4; Test type: Superiority; p = 0.963, Cochran-Mantel-Haenszel; Absolute Difference = -2.2, 95% CI 2-sided [-32.1 to 27.8]

6. Secondary Outcome: SRI-4 Response With a Sustained Reduction of OCS Dose to ≤ 10 mg/Day and ≤ Day 1 Dose During Week 36 Through 48 in Patients With High vs. Low Plasmablast Signature Levels
Description: as for outcome 5
Time Frame: Week 48
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID
Number analyzed (Participants) | 24 | 24 | 25
Percentage of Participants
  Plasmablast Signature Level Q1: number analyzed (Participants) | 24 | 21 | 20
  Plasmablast Signature Level Q1 | 33.3 | 52.4 | 40.0
  Plasmablast Signature Level Q2: number analyzed (Participants) | 22 | 24 | 19
  Plasmablast Signature Level Q2 | 54.5 | 54.2 | 57.9
  Plasmablast Signature Level Q3: number analyzed (Participants) | 19 | 21 | 25
  Plasmablast Signature Level Q3 | 36.8 | 52.4 | 44.0
  Plasmablast Signature Level Q4: number analyzed (Participants) | 20 | 21 | 23
  Plasmablast Signature Level Q4 | 45.0 | 42.9 | 39.1
Statistical Analysis 1: Comparison: Placebo vs GDC-0853 (150mg) QD; Plasmablast Signature Level Q1; Test type: Superiority; p = 0.189, Cochran-Mantel-Haenszel; Absolute Difference = 19.0, 95% CI 2-sided [-9.4 to 47.5]
Statistical Analysis 2: Comparison: Placebo vs GDC-0853 (200mg) BID; Plasmablast Signature Level Q1; Test type: Superiority; p = 0.909, Cochran-Mantel-Haenszel; Absolute Difference = 6.7, 95% CI 2-sided [-21.9 to 35.2]
Statistical Analysis 3: Comparison: Placebo vs GDC-0853 (150mg) QD; Plasmablast Signature Level Q2; Test type: Superiority; p = 0.500, Cochran-Mantel-Haenszel; Absolute Difference = -0.4, 95% CI 2-sided [-29.2 to 28.4]
Statistical Analysis 4: Comparison: Placebo vs GDC-0853 (200mg) BID; Plasmablast Signature Level Q2; Test type: Superiority; p = 0.234, Cochran-Mantel-Haenszel; Absolute Difference = 3.3, 95% CI 2-sided [-27.1 to 33.8]
Statistical Analysis 5: Comparison: Placebo vs GDC-0853 (150mg) QD; Plasmablast Signature Level Q3; Test type: Superiority; p = 0.364, Cochran-Mantel-Haenszel; Absolute Difference = 15.5, 95% CI 2-sided [-14.9 to 46]
Statistical Analysis 6: Comparison: Placebo vs GDC-0853 (200mg) BID; Plasmablast Signature Level Q3; Test type: Superiority; p = 0.310, Cochran-Mantel-Haenszel; Absolute Difference = 7.2, 95% CI 2-sided [-22 to 36.3]
Statistical Analysis 7: Comparison: Placebo vs GDC-0853 (150mg) QD; Plasmablast Signature Level Q4; Test type: Superiority; p = 0.922, Cochran-Mantel-Haenszel; Absolute Difference = -2.1, 95% CI 2-sided [-32.5 to 28.2]
Statistical Analysis 8: Comparison: Placebo vs GDC-0853 (200mg) BID; Plasmablast Signature Level Q4; Test type: Superiority; p = 0.701, Cochran-Mantel-Haenszel; Absolute Difference = -5.9, 95% CI 2-sided [-35.4 to 23.7]

7. Secondary Outcome: SRI-6 Response at Week 24 and 48
Description: The Systemic Lupus Erythematosus Responder Index (SRI)-6 measures reduction in SLE disease activity and is a composite measure that includes the SLE Disease Activity Index (SLEDAI-2K), British Isles Lupus Activity Group (BILAG) 2004 and Physician Global Assessment. It is defined as: 1) Reduction of ≥6 points from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score; 2) no new British Isles Lupus Assessment Group (BILAG) A or no more than 1 new BILAG B disease activity scores and 3) no worsening (defined as an increase of ≥0.3 points [10 mm] from baseline) in the Physician's Global Assessment of Disease Activity. The score range is from 0 to 100, with higher scores indicating greater disease activity.
Time Frame: Week 24, 48
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID
Number analyzed (Participants) | 86 | 87 | 87
Percentage of Participants
  Week 24 | 31.4 | 34.5 | 33.3
  Week 48 | 27.9 | 39.1 | 35.6
Statistical Analysis 1: Comparison: Placebo vs GDC-0853 (150mg) QD; Week 24; Test type: Superiority; p = 0.692, Cochran-Mantel-Haenszel; Absolute Difference = 3.1, 95% CI 2-sided [-10.9 to 17.1]
Statistical Analysis 2: Comparison: Placebo vs GDC-0853 (200mg) BID; Week 24; Test type: Superiority; p = 0.871, Cochran-Mantel-Haenszel; Absolute Difference = 1.9, 95% CI 2-sided [-12 to 15.9]
Statistical Analysis 3: Comparison: Placebo vs GDC-0853 (150mg) QD; Week 48; Test type: Superiority; p = 0.105, Cochran-Mantel-Haenszel; Absolute Difference = 11.2, 95% CI 2-sided [-2.8 to 25.1]
Statistical Analysis 4: Comparison: Placebo vs GDC-0853 (200mg) BID; Week 48; Test type: Superiority; p = 0.286, Cochran-Mantel-Haenszel; Absolute Difference = 7.7, 95% CI 2-sided [-6.1 to 21.6]

8. Secondary Outcome: BILAG-based Composite Lupus Assessment (BICLA) Response at Week 24 and 48
Description: The BICLA is a composite index that is defined as follows: [1] At least one gradation of improvement in baseline BILAG scores in all body systems with moderate or severe disease activity at entry (e.g., all A (severe disease) scores falling to B (moderate), C (mild), or D (no activity) and all B scores falling to C or D; [2] No new BILAG A or more than one new BILAG B scores; [3] No worsening of total SLEDAI-2K score from baseline; [4] No significant deterioration (=<10%) in physician's global assessment and [5] No treatment failure (initiation of non-protocol treatment).
Time Frame: Week 24, 48
Population: The BICLA-evaluable population was defined as all all ITT participants who had at least one body system with moderate or severe disease activity at baseline as determined by BILAG-2004, i.e., at least one BILAG domain was scored as A or B at baseline.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID
Number analyzed (Participants) | 80 | 85 | 83
Percentage of Participants
  Week 24 | 47.5 | 45.9 | 44.6
  Week 48 | 41.2 | 52.9 | 42.2
Statistical Analysis 1: Comparison: Placebo vs GDC-0853 (150mg) QD; Week 24; Test type: Superiority; p = 0.936, Cochran-Mantel-Haenszel; Absolute Difference = -1.6, 95% CI 2-sided [-16.8 to 13.6]
Statistical Analysis 2: Comparison: Placebo vs GDC-0853 (200mg) BID; Week 24; Test type: Superiority; p = 0.683, Cochran-Mantel-Haenszel; Absolute Difference = -2.9, 95% CI 2-sided [-18.2 to 12.4]
Statistical Analysis 3: Comparison: Placebo vs GDC-0853 (150mg) QD; Week 48; Test type: Superiority; p = 0.086, Cochran-Mantel-Haenszel; Absolute Difference = 11.7, 95% CI 2-sided [-3.4 to 26.8]
Statistical Analysis 4: Comparison: Placebo vs GDC-0853 (200mg) BID; Week 48; Test type: Superiority; p = 0.879, Cochran-Mantel-Haenszel; Absolute Difference = 0.9, 95% CI 2-sided [-14.2 to 16.1]

9. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An Adverse Event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to 8 weeks after the last dose of study drug (up to Week 56).
Population: The Safety-evaluable population was defined as all participants who received at least one dose of study medication. One participant in the Placebo arm was inadvertently dosed with GDC-0853 for a period of 27 days and was classified as part of the GDC-0853 (200mg) BID arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID
Number analyzed (Participants) | 84 | 87 | 88
Percentage of Participants | 76.2 | 88.5 | 78.4

10. Secondary Outcome: Plasma Concentrations of Fenebrutinib at Specified Timepoints
Description: The PK analyses includes tabulation of plasma concentration data and summarisation of plasma concentrations by visits with participants grouped according to treatment received. Descriptive summary statistics for the Arithmetic Mean and Standard Deviation are presented below.
Time Frame: Baseline (Pre-dose), Week 24 (Pre-dose and Post-dose) and Week 48 (Pre-dose)
Population: The PK-evaluable population was defined as all participants who received at least one dose of fenebrutinib (GDC-0853) and had at least 1 evaluable post-dose PK sample. Data presented below is only for participants that were included in the actual analysis with detectable concentrations at the specified timepoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID
Number analyzed (Participants) | 87 | 86
ng/mL
  Week 0 (Pre-dose) | NA (NA) — No Drug was administered at this timepoint and so there were no detectable concentrations. | NA (NA) — No Drug was administered at this timepoint and so there were no detectable concentrations.
  Week 24 (Pre-dose): number analyzed (Participants) | 67 | 68
  Week 24 (Pre-dose) | 41.9 (62.4) | 180 (121)
  Week 24 (2hr Post-dose): number analyzed (Participants) | 66 | 67
  Week 24 (2hr Post-dose) | 331 (226) | 612 (353)
  Week 24 (4-6hr Post-dose): number analyzed (Participants) | 65 | 66
  Week 24 (4-6hr Post-dose) | 215 (131) | 414 (187)
  Week 24 (8-10hr Post-dose): number analyzed (Participants) | 11 | 7
  Week 24 (8-10hr Post-dose) | 120 (111) | 233 (145)
  Week 48 (Pre-dose): number analyzed (Participants) | 64 | 64
  Week 48 (Pre-dose) | 25.5 (28.1) | 137 (133)

ADVERSE EVENTS:
Time Frame: Baseline up to 8 weeks after the last dose of study drug (up to Week 56).
Description: The Safety Population was defined as all participants who received at least one dose of study medication. One participant in the Placebo arm was inadvertently dosed with GDC-0853 for a period of 27 days and was classified as part of the GDC-0853 (200mg) BID arm. AEs that were entered into the database at the time of the database lock were included in the AE analysis.
Arm/Group | Placebo | GDC-0853 (150mg) QD | GDC-0853 (200mg) BID
All-Cause Mortality (participants affected / at risk) | 2/84 | 1/87 | 0/88
Serious Adverse Events (participants affected / at risk) | 9/84 | 4/87 | 12/88
Other Adverse Events (participants affected / at risk) | 42/84 | 54/87 | 51/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=84) | GDC-0853 (150mg) QD (N=87) | GDC-0853 (200mg) BID (N=88)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
MYOCARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 1 (1)
EPSTEIN-BARR VIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INFECTED SKIN ULCER (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OSTEOMYELITIS CHRONIC (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
CHEST WALL HAEMATOMA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
CERVIX CARCINOMA STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=84) | GDC-0853 (150mg) QD (N=87) | GDC-0853 (200mg) BID (N=88)
LYMPHOPENIA (Blood and lymphatic system disorders) | 6 (6) | 2 (2) | 10 (12)
NEUTROPENIA (Blood and lymphatic system disorders) | 4 (5) | 5 (5) | 6 (6)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 2 (2) | 5 (7)
DIARRHOEA (Gastrointestinal disorders) | 6 (6) | 5 (8) | 5 (6)
NAUSEA (Gastrointestinal disorders) | 7 (7) | 4 (4) | 7 (7)
BRONCHITIS (Infections and infestations) | 6 (7) | 6 (6) | 7 (9)
GASTROENTERITIS (Infections and infestations) | 5 (7) | 2 (2) | 2 (2)
INFLUENZA (Infections and infestations) | 5 (8) | 5 (5) | 5 (5)
NASOPHARYNGITIS (Infections and infestations) | 5 (6) | 8 (12) | 6 (6)
SINUSITIS (Infections and infestations) | 3 (3) | 2 (2) | 5 (5)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (7) | 9 (10) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 9 (11) | 17 (21) | 11 (15)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 5 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (3) | 8 (9) | 4 (4)
HEADACHE (Nervous system disorders) | 9 (10) | 3 (4) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT02908100/Prot_SAP_000.pdf